CLINICAL TRIAL: NCT00669877
Title: Rituximab and Hyper-CVAD (Cyclophosphamide, Vincristine, Adriamycin, and Dexamethasone) for Burkitt's and Burkitt's -Like Leukemia/Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID02-229; NCI-2010-01455 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2008-04-28; First posted 2008-05-01 (Estimated); Results first posted 2018-05-16 (Actual); Last update posted 2018-05-16 (Actual); Status verified 2018-04

CONDITIONS: Burkitt's Lymphoma; Burkitt'S-like Lymphoma
Keywords: Burkitt's Lymphoma; Burkitt's Like Lymphoma; Leukemia; Hyper-CVAD; Rituximab; Methotrexate; Cytarabine
MeSH Terms: conditions — Burkitt Lymphoma; Leukemia | interventions — Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Dexamethasone; Calcium Dobesilate; Granulocyte Colony-Stimulating Factor; Filgrastim; Cytarabine; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hyper-CVAD (Experimental): Hyper-CVAD (odd courses) alternated with high-dose methotrexate + cytarabine (even courses) every 21 days or later to allow for myelosuppression recovery, for total of 8 courses. Rituximab 375 mg/m2 days 1 +/- 2 days and 11 +/- 2 days for the odd courses of therapy, and days 1 +/- 2 days and 8 +/- 2 days for the even courses of therapy, first 4 courses. Cyclophosphamide 300 mg/m2 IV over 3 hours every 12 hours x 6 doses days 1, 2, 3. Doxorubicin 50 mg/m2 IV over 2-24 hours via CVC on day 4 after last dose of cyclophosphamide given (odd courses). Vincristine 2 mg IV on day 4 +/- 2 days and day 11 +/- 2 days (odd courses). Dexamethasone 40 mg IV or by mouth (P.O.) daily days 1-4 +/- 2 days and days 11-14 +/- 2 days (odd courses). G-CSF 10 mg/kg/day (rounded) until neutrophil recovery 1 x 10^9/L or higher can be substituted or can be added to pegfilgrastim if neutrophils have not recovered to 1 x 10^9/L by day 21.
  Interventions: Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Dexamethasone; Drug: G-CSF; Drug: Cytarabine; Drug: Methotrexate

INTERVENTIONS:
Drug: Rituximab — 375 mg/m2 IV days 1 +/- 2 days and 11 +/- 2 days for the odd courses of therapy, and days 1 +/- 2 days and 8 +/- 2 days for the even courses of therapy, first 4 courses.
  Other Names: Rituxan
Drug: Cyclophosphamide — 300 mg/m2 IV over 3 hours every 12 hours x 6 doses days 1, 2, 3 (total dose 1800 mg/m2) starting after rituximab completed (odd courses).
  Other Names: Cytoxan; Neosar
Drug: Doxorubicin — 50 mg/m2 IV over 2-24 hours via CVC on day 4 after last dose of cyclophosphamide given (odd courses).
  Other Names: Adriamycin; Rubex
Drug: Vincristine — 2 mg IV on day 4 +/- 2 days and day 11 +/- 2 days (odd courses)
  Other Names: Oncovin; Vincasar Pfs
Drug: Dexamethasone — 40mg IV or by mouth (P.O.) daily days 1-4 +/- 2 days and days 11-14 +/- 2 days (odd courses)
  Other Names: Decadron
Drug: G-CSF — 10 mcg/kg
  Other Names: Filgrastim; Neupogen
Drug: Cytarabine — 100 mg intrathecal day 7 +/- 2 days (odd courses); 3 gm/m2 IV over 2 hours every 12 hours for 4 doses on days 2, 3 (even courses).
  Other Names: Ara-C; Cytosar; DepoCyt; Cytosine Arabinosine Hydrochloride
Drug: Methotrexate — 200 mg/m2 IV over 2 hrs followed by 800 mg/m2 over 22 hrs on day 1 after the completion of Rituximab.
  Other Names: Rheumatrex; Methotrexate Sodium, MTX

SUMMARY:
The goal of this clinical research study is to learn if intensive chemotherapy given over 6 months can help to control or cure Burkitt's leukemia, Burkitt's lymphoma, or small non-cleaved cell B-cell leukemia or lymphoma. Another goal is to see how well this treatment works when given with Rituximab. The safety of the combined treatment will also be studied.

DETAILED DESCRIPTION:
The hyper-CVAD regimen is a combination of chemotherapy drugs including cyclophosphamide, vincristine, Adriamycin, and dexamethasone given together to for one "course" of treatment. This alternates with a course or combination of the chemotherapy drugs methotrexate and cytarabine. Rituximab is a protein (monoclonal antibody) that attaches to the surface of the leukemia or lymphoma cells which have a marker called cluster of differentiation antigen 20 (CD20).

During treatment, participants will have a physical exam and give blood samples (about 1 tablespoon each) at least twice a week. After two courses of chemotherapy, the tests done before treatment will be repeated to check for response. In patients with leukemia, a bone marrow sample will be repeated 2 and 3 weeks from the beginning of treatment to check the response.

All participants in this study will receive 2 kinds of chemotherapy courses for a total of 8 courses. Chemotherapy courses will be given through a large vein by a central venous catheter (a plastic tube usually placed under the collarbone).

In Course 1 (odd course), participants will receive rituximab by vein over 6 hours on Days 1 and 11. Participants will receive the drugs acetaminophen (Tylenol) and diphenhydramine hydrochloride (Benadryl) 30-60 minutes before each dose of rituximab. This will be done to lessen the risk of fever, chills, and allergic reactions. Usually, the first dose of rituximab requires about 6 hours to complete.

Participants will then receive cyclophosphamide by vein over 2-3 hours every 12 hours for a total of 6 doses, given over 3 days (Days 1, 2, and 3). Adriamycin will be given by vein over 24 hours on Day 4. Vincristine will be given by vein over 15 to 30 minutes on Days 4 and 11 along with dexamethasone by mouth or by vein on Days 1-4 and 11-14.

Participants will also receive pegfilgrastim or G-CSF (growth stimulating colony factor) to help with rapid recovery of the normal bone marrow starting after each course of chemotherapy is finished. Pegfilgrastim is injected under the skin within 72 hours of completion of each cycle of chemotherapy. G-CSF is given by injections by vein or under the skin until the blood counts recover.

Treatment to the brain will be given inside the spinal fluid with cytarabine and methotrexate about Days 2 and 7 of the course to help prevent the leukemia from developing there.

For patients 60 years or older, the first course will be given in a protective isolation room to decrease the risk of infection(s).

In Course 2 (even course), participants will receive rituximab by infusion over about 4 hours on Days 1 and 8. They will receive methotrexate by infusion over 24 hours on the first day, and cytarabine in a high dose over 2 hours every 12 hours for 4 doses (Days 2 and 3). Citrovorum factor (leucovorin) will be given by vein or by mouth for 2-3 days (Day 2 and on) to decrease the risk of side effects of methotrexate. G-CSF will be given as in Course 1 (after the chemotherapy is finished). The treatment to the brain inside the spinal fluid will be given as in course 1 on days 2 and 7.

After two courses of therapy, the response to the treatment will be checked. If the leukemia or lymphoma is responding, the therapy will be continued for a total of 8 courses over 6 months. Therapy will be stopped if the leukemia or lymphoma starts to get worse.

An Ommaya reservoir may also be placed surgically as a route to treat leukemia in the brain or to decrease the risk of leukemia in patients who have difficulty with the spinal treatments. An Ommaya reservoir is a tube inserted under the skin of the scalp that enters into the spinal fluid cavity of the brain.

This is an investigational study. All drugs in this study are commercially available. Their use together in this study is investigational. About 70 patients or more will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Burkitt's or Burkitt-like leukemia and/or lymphoma, either previously untreated, previously treated (may be in CR or with active disease after 1-2 courses of chemotherapy), or HIV-related.
2. All ages are eligible.
3. Zubrod performance status < 3 (ECOG Scale, Appendix A).
4. Adequate liver function (bilirubin < 3.0 mg/dL, unless considered due to tumor), and renal function (creatinine < 3.0 mg/dL, unless considered due to tumor).
5. Signed informed consent.

Exclusion Criteria:

1) N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2002-08; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan O'Brien, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: August 15, 2002 to August 28, 2012. All recruitment done at The University of Texas (UT) MD Anderson Cancer Center.
Period: Overall Study
Arm/Group | Hyper-CVAD
Started | 56
Completed | 52
Not Completed | 4
Not completed — Disease Progression/Death | 4

BASELINE CHARACTERISTICS:
Arm/Group | Hyper-CVAD
Number analyzed (Participants) | 56
Age, Continuous [Median (Full Range); unit: years] | 41 [17 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 37
Region of Enrollment [Number; unit: participants]
  United States | 56

OUTCOME MEASURES:

1. Primary Outcome: Complete Remission Rate: Percentage of Participants With Complete Remission (CR)
Description: Complete Remission (CR) was defined as the presence of 5% or less blasts in the bone marrow, with a granulocyte count ≥1.0 × 10^9/L, a platelet count ≥100 × 10^9/L, and no extramedullary disease. Complete recovery except platelets (CRp) was defined as for CR, except for recovery of platelet count to <100 × 10^9/L. Partial remission (PR) was defined as a bone marrow with >5% and <25% blasts with a granulocyte count of ≥1.0 × 109/L and a platelet count of ≥100 × 10^9/L. Relapse was defined by recurrence of more than 5% lymphoblasts in the bone marrow aspirate or by the presence of extramedullary disease after achieving CR.
Time Frame: After two 21-day courses, response to treatment checked for Complete Remission (CR)
Population: Of fifty-six registered, nine participants entered the study with CR therefore were not evaluable for response.
Measure: Number; unit: percentage of participants
Arm/Group | Hyper-CVAD
Number analyzed (Participants) | 47
percentage of participants | 85

2. Other Pre Specified Outcome: Overall Response Rate: Percentage of Participants With Complete Remission (CR) or Partial Remission (PR)
Description: as for outcome 1
Time Frame: After two 21-day courses, response to treatment checked for Complete Remission (CR)
Population: Of fifty-six registered, nine participants entered the study with CR therefore were not evaluable for response.
Measure: Number; unit: percentage of participants
Arm/Group | Hyper-CVAD
Number analyzed (Participants) | 47
percentage of participants | 89

ADVERSE EVENTS:
Time Frame: Adverse events collected through alternating treatment cycles, every 21 days or later to allow for recovery from myelosuppression, for a total of 8 courses or a total of 24 weeks.
Arm/Group | Hyper-CVAD
Serious Adverse Events (participants affected / at risk) | 27/56
Other Adverse Events (participants affected / at risk) | 47/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Hyper-CVAD (N=56)
Febrile Neutropenia (Blood and lymphatic system disorders) | 27
Urinary Infection (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 5
Cholecystitis (Hepatobiliary disorders) | 1
Cytomegalovirus retinitis (CMV retinitis) (Eye disorders) | 1
Hemorrhage with Thrombopenia (Blood and lymphatic system disorders) | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
Altered Mental Status (Psychiatric disorders) | 1
Arrhythmia (Cardiac disorders) | 1
Cardiac Ischemia (Cardiac disorders) | 1
Death (General disorders) | 3
Fever without neutropenia (Investigations) | 3
Fracture, Hip (Injury, poisoning and procedural complications) | 1
Hemorrhage, Central Nervous System (Nervous system disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hypotension (Cardiac disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Infection with neutropenia (Infections and infestations) | 7
Infection with normal ANC (Infections and infestations) | 1
Infection without neutropenia (Infections and infestations) | 3
Infection, Blood (Infections and infestations) | 1
Infection, wound (Infections and infestations) | 1
Neuropathy (Nervous system disorders) | 1
Non-Neutropenic Fever (Investigations) | 3
Perforation, GI Small Bowel (Gastrointestinal disorders) | 1
Renal Failure (Renal and urinary disorders) | 1
Seizures (Nervous system disorders) | 1
Thrombosis (Vascular disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Hyper-CVAD (N=56)
Bacterial Infection (Infections and infestations) | 16
Fever, Unknown Origin (General disorders) | 24
Pneumonia, Unknown Pathogen (Infections and infestations) | 16
Bacterial Pneumonia (Infections and infestations) | 4
Viral Infection (Infections and infestations) | 4
Non-specified infections (Infections and infestations) | 4
Hypokalemia (Metabolism and nutrition disorders) | 1
Elevated Alkaline phosphatase (ALT) (Investigations) | 1
Hemorrhage (General disorders) | 1
Acute Renal Failure (Renal and urinary disorders) | 1
Mucositis (Gastrointestinal disorders) | 1
Peripheral Neuropathy (Nervous system disorders) | 1
Vomiting (General disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes